CLINICAL TRIAL: NCT00213733
Title: Research of Molecular Markers for Diagnosis and/or Prognosis in Lymph Node Metastasis of Resected Non-small Cell Lung Cancer
Brief Title: Molecular Assessment of Lymph Nodes in Patients With Resected (Stage I to IIIA) Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Emmanuel LAVOUE, Directeur Adjoint de la DRCI, University Hospital, Strasbourg, France
Other Study IDs: 3207
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Lung Cancer
Keywords: Lung cancer patients; non-small cell lung cancer; molecular marker; lymph node completed resected; Lung cancer samples and paired lymph node resected
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This is a prospective study of surgically resected samples and lymph nodes of lung cancer patients. For histopathologically positive lymph nodes from a complete resection, the investigators would like to analyse tumor tissue by allelotyping and comparing these results with those observed in the primary lung tumor to establish a cartography of molecular alteration in resected lung cancer. For non histopathologically positive lymph nodes, the investigators would like to research the presence (or not) of micrometastasis by allele-specific PCR (polymerase chain reaction).

DETAILED DESCRIPTION:
Genetic: It is a prospective study during two years with three years for follow-up. No control group is recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resectable non-small cell lung cancer (stage I to IIIA), with a complete resection of the tumor and paired lymph nodes.
* Informed consent is required.

Exclusion Criteria:

* Another cancer
* Chemotherapy before surgical treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with resectable non-small cell lung cancer (stage I to IIIA), with a complete resection of the tumor and paired lymph nodes
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2004-06; Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michèle BEAU-FALLER, MD, Principal Investigator — Laboratoire de Biochimie et de Biologie Moléculaire, Hôpital de Hautepierre
Locations (5):
- France (5):
  - Service de Chirurgie Thoracique, Hôpital Civil, Strasbourg
  - Service de Pneumologie, Hôpital Lyautey, Strasbourg
  - Laboratoire de Biochimie et de Biologie Moléculaire, Hôpital de Hautepierre, Strasbourg
  - Service d'Anatomie Pathologique, Hôpital de Hautepierre, Strasbourg
  - Service de Pneumologie, Hôpital de Hautepierre, Strasbourg